CLINICAL TRIAL: NCT00002320
Title: A Randomized, Double-Blind Multicenter Trial to Compare the Safety and Efficacy of Lamivudine (3TC; GR109714X) Monotherapy Versus Zidovudine (AZT) Monotherapy Versus 3TC Administered With AZT in the Treatment of HIV-1 Infected Patients Who Are AZT Naive (< 4 Weeks) With CD4 Cell Counts of 200-500 Cells/mm3
Brief Title: A Comparison of Lamivudine and Zidovudine, Used Alone and Together, in HIV-Infected Patients Who Have Not Used Zidovudine in the Past
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 129B; NUCA 3001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-12-12 (Estimated); Status verified 1994-05

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To evaluate the safety and efficacy of high-dose lamivudine (3TC) alone versus zidovudine (AZT) alone versus 3TC at high and low doses in combination with AZT in HIV-1 infected patients.

PER 02/27/95 AMENDMENT: To evaluate the efficacy and safety of both blinded and open-label combination therapy.

DETAILED DESCRIPTION:
Patients are randomized to one of four treatment arms: 3TC alone, AZT alone, low-dose 3TC plus AZT, or high-dose 3TC plus AZT. Patients receive treatment for 32 weeks, with possible extension to 52 weeks.

PER 02/27/95 AMENDMENT: Patients may continue therapy on AZT and low-dose 3TC on an open-label basis. Open-label therapy continues with follow-up every 8 weeks until intolerable toxicity occurs or study terminates.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity.
* CD4 count 200-500 cells/mm3.
* AZT naive status (<= 4 weeks of prior AZT).

Exclusion Criteria

Patients with the following prior condition are excluded:

History of intolerance to AZT.

Prior Medication:

Excluded:

* More than 4 weeks of prior AZT.
* Any prior antiretroviral treatment other than AZT.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320

CONTACTS AND LOCATIONS:
Locations (22):
- United States (18):
  - Combat Group, Los Angeles, California
  - San Diego Community Research Group, San Diego, California
  - Pacific Oaks Med Group, Sherman Oaks, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Louisiana Cardiovascular Research Ctr, New Orleans, Louisiana
  - CRI of New England, Brookline, Massachusetts
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Univ of North Carolina School of Medicine, Chapel Hill, North Carolina
  - Med College of Ohio, Toledo, Ohio
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Mem Hosp of Rhode Island, Pawtucket, Rhode Island
  - Central Texas Med Foundation, Austin, Texas
  - Nicholaos Bellos, Dallas, Texas
  - Richmond AIDS Consortium, Richmond, Virginia
  - Wisconsin Community - Based Research Consortium, Milwaukee, Wisconsin
- Canada (3):
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto Hosp, Toronto, Ontario
  - Montreal Gen Hosp, Montreal, Quebec
- Advance Community Health Services Inc, Santurce, Puerto Rico

REFERENCES:
- [Background] Eron JJ Jr. The treatment of antiretroviral-naive subjects with the 3TC/zidovudine combination: a review of North American (NUCA 3001) and European (NUCB 3001) trials. AIDS. 1996 Dec;10 Suppl 5:S11-9. doi: 10.1097/00002030-199612005-00003. PMID 9030391
- [Background] Kuritzkes DR, Quinn JB, Benoit SL, Shugarts DL, Griffin A, Bakhtiari M, Poticha D, Eron JJ, Fallon MA, Rubin M. Drug resistance and virologic response in NUCA 3001, a randomized trial of lamivudine (3TC) versus zidovudine (ZDV) versus ZDV plus 3TC in previously untreated patients. AIDS. 1996 Aug;10(9):975-81. doi: 10.1097/00002030-199610090-00007. PMID 8853730